CLINICAL TRIAL: NCT02118220
Title: Effects of Anesthesia on Pediatric Surgical Patients With a History of Concussion - Phase I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Lynne Ferrari, Chief, Perioperative Anesthesia, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-P00011568
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Post Concussion Symptoms
MeSH Terms: conditions — Post-Concussion Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Concussion Questionnaire (Other): The questionnaire is specifically designed to elicit occurrence and symptoms of a concussion. If the patient answers yes to question 2a, which asks "At the time of the injury do you recall a blow to the head, neck, face or body that resulted in sustained symptoms of concussion (e.g., headache, dizziness, confusion, nausea, vomiting, etc.)?", the research team will administer the 22 item self-reporting symptom scale in the above mentioned SCAT3. The responses obtained from the questionnaire will be used to determine the incidence of symptomatic concussions, either known or unrecognized, in pediatric patients sustaining an orthopedic injury requiring surgical repair.
  Interventions: Other: Concussion Questionnaire

INTERVENTIONS:
Other: Concussion Questionnaire

SUMMARY:
The purpose of this research study is to determine the number of children who have symptoms of a concussion at the time they are scheduled for orthopedic surgery at Boston Children's Hospital. It is currently unknown if anesthesia affects a child with a previously diagnosed concussion. This study is the first phase of a two-part study looking at the effects of anesthesia in children undergoing orthopedic surgery with a previous concussion. Currently, the decision to continue with surgery in patients with a diagnosed concussion is based on clinical judgment by the patients.

DETAILED DESCRIPTION:
Phase I's specific aim is to estimate the incidence of symptomatic concussion in the pediatric orthopedic surgical population.

The first phase of this study requires a member of the research team to administer a paper questionnaire to all eligible, consented orthopedic surgery patients in either the Pre-operative Clinic or in the Day Surgery Unit over a period of four months. The research member will only approach adolescents that are scheduled for repair of orthopedic traumatic injury as defined in the inclusion criteria. The questionnaire is specifically designed to elicit occurrence and symptoms of a concussion. If the patient answers yes to question 2a, which asks "At the time of the injury do you recall a blow to the head, neck, face or body that resulted in sustained symptoms of concussion (e.g., headache, dizziness, confusion, nausea, vomiting, etc.)?", the research team will administer the 22 item self-reporting symptom scale in the above mentioned SCAT3. The responses obtained from the questionnaire will be used to determine the incidence of symptomatic concussions, either known or unrecognized, in pediatric patients sustaining an orthopedic injury requiring surgical repair. If the participant scores higher than a 0 on the SCAT3 the results will be conveyed to the surgeon prior to the start of the scheduled surgical procedure. A copy of the completed SCAT3 will also be placed in the medical record. The decision to continue with surgery and need to possibly refer the patient to the Boston Children's Hospital Sports Concussion Clinic after the SCAT3 will remain at the surgeon's discretion.

Information will be gathered from the questionnaire and the SCAT3, then entered into the REDcap database under a de-identified subject number.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 5-21 years of age presenting for repair of orthopedic traumatic injury. Orthopedic traumatic injury will be defined as any traumatic injury resulting from a fall, collision (struck by or struck against), vehicle accident, assault or bike-related injury or fracture.

Exclusion Criteria:

Patients who do not speak English as their first language, or who are unable to respond to the survey's questions on their own will be excluded from study participation.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2014-05; Primary Completion 2015-04 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Estimate the incidence of symptomatic concussion in the pediatric orthopedic surgical population. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Ferrari, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Gessel LM, Fields SK, Collins CL, Dick RW, Comstock RD. Concussions among United States high school and collegiate athletes. J Athl Train. 2007 Oct-Dec;42(4):495-503. PMID 18174937
- [Background] SCAT3. Br J Sports Med. 2013 Apr;47(5):259. No abstract available. PMID 23479480
- [Background] Child SCAT3. Br J Sports Med. 2013 Apr;47(5):263. No abstract available. PMID 23479481
- [Background] McCrea M, Hammeke T, Olsen G, Leo P, Guskiewicz K. Unreported concussion in high school football players: implications for prevention. Clin J Sport Med. 2004 Jan;14(1):13-7. doi: 10.1097/00042752-200401000-00003. PMID 14712161
- [Background] Meehan WP 3rd, Bachur RG. Sport-related concussion. Pediatrics. 2009 Jan;123(1):114-23. doi: 10.1542/peds.2008-0309. PMID 19117869
- [Background] Zhou Y, Kierans A, Kenul D, Ge Y, Rath J, Reaume J, Grossman RI, Lui YW. Mild traumatic brain injury: longitudinal regional brain volume changes. Radiology. 2013 Jun;267(3):880-90. doi: 10.1148/radiol.13122542. Epub 2013 Mar 12. PMID 23481161